CLINICAL TRIAL: NCT01889160
Title: A Phase I Single-blind, Randomised, Placebo-controlled, Single-centre Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Oral AZD4721 Solution After Single Ascending Doses, and to Compare the Oral Bioavailability of Single Doses of Solution and Suspension in Healthy Subjects
Brief Title: Study to Investigate the Safety Profile of AZD4721 After Single Doses at Different Dose Levels
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: D5200C00001
Record Dates: First submitted 2013-06-24; First posted 2013-06-28 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Safety,Plasma AUC and Cmax, Plasma AUC 0-t, t1/2λz, and Tmax
Keywords: Healthy volunteers, Phase 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part A Active (Experimental): AZD4721 Solution
  Interventions: Drug: AZD4721 Solution
- Part A Placebo (Placebo Comparator): Placebo for AZD4721
  Interventions: Drug: AZD4721 Placebo
- Part B solution (Experimental): AZD4721 Solution
  Interventions: Drug: AZD4721 Solution
- Part B Suspension (Active Comparator): AZD4721 Suspension
  Interventions: Drug: AZD4721 Suspension

INTERVENTIONS:
Drug: AZD4721 Solution — 1-9 mg/mL liquid solution
  Arms: Part A Active; Part B solution
Drug: AZD4721 Placebo — Liquid solution
  Arms: Part A Placebo
Drug: AZD4721 Suspension — 9 mg/g liquid suspension
  Arms: Part B Suspension

SUMMARY:
Study to investigate the safety profile of AZD4721 after single doses at different dose levels

DETAILED DESCRIPTION:
A study to investigate safety and tolerability of single ascending doses of AZD4721 given to healthy volunteers. Including a bioequivalence part to compare a solution of AZD4721 with a suspension.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and/or female Caucasian (neither Black/African American nor Japanese) volunteers aged 18-50 years. ("Healthy" is as determined by medical history and physical examination, clinical laboratory parameters, and ECG )
2. Females must have a negative pregnancy test at screening and on admission to the unit, must not be lactating and must be of nonchildbearing potential
3. Volunteers should have a BMI between 18 and 30 kg/m2 (inclusive) and weigh at least 50 kg and no more than 100 kg (inclusive).

Exclusion Criteria:

1. History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate
2. Current smokers or those who have smoked or used nicotine products within the previous 3 months

2.Clinically significant lower respiratory tract infection not resolved within 4 weeks prior to Visit 1, as determined by the Investigator

4. Other latent or chronic infections (eg, recurrent sinusitis, genital or ocular herpes, urinary tract infection) or at risk of infection (surgery, trauma, or significant infection) in previous 90 days, or history of skin abscesses within the previous

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Description of the safety profile in terms of Adverse events; blood pressure, heart rate and body temperature; electrocardiograms; clinical chemistry; haematology assessments, including serial blood neutrophil count | From Screening to follow up ( maximum 7 weeks)

SECONDARY OUTCOMES:
Description of the pharmacokinetic(PK) profile for in terms of: observed maximum plasma concentration (Cmax), time to reach maximum plasma concentration (tmax), terminal rate constant (λz), terminal half-life (t½ z). | Sample taken predose, 1, 3, 5, 7, 9, 13, 18, 24, 36, 48, 72, 96, 144, 216 hours postdose
Description of the pharmacokinetic(PK) profile for in terms of: area under the plasma concentration-time curve from time zero to 24 hours after dosing (AUC(0-24)), from time zero to the time of last quantifiable concentration (AUC(0 last)) | Sample taken predose, 1, 3, 5, 7, 9, 13, 18, 24, 36, 48, 72, 96, 144, 216 hours postdose
Description of the pharmacokinetic(PK) profile for in terms of from time zero extrapolated to infinity (AUC), apparent clearance for parent drug estimated as dose divided by AUC (CL/F; AZD4721 only) | Sample taken predose, 1, 3, 5, 7, 9, 13, 18, 24, 36, 48, 72, 96, 144, 216 hours postdose
Description of the pharmacokinetic(PK) profile in terms of apparent volume of distribution during terminal phase (Vz/F; AZD4721 only), mean residence time (MRT, AZD4721 only), lag-time (T-lag, AZD4721 only), dose-normalized AUC (AUC/D) and Cmax (Cmax/D) | Sample taken predose, 1, 3, 5, 7, 9, 13, 18, 24, 36, 48, 72, 96, 144, 216 hours postdose
Description of the pharmacokinetic(PK) profile for in terms of effective half-life (t½(eff)), time of last quantifiable concentration (tlast), predicted accumulation ratio (Rac,pred) | Sample taken predose, 1, 3, 5, 7, 9, 13, 18, 24, 36, 48, 72, 96, 144, 216 hours postdose
Description of the pharmacokinetic(PK) profile for in terms of the time interval and number of data points included in the log-linear regression to determine terminal half-life (z,Interval and z,N) | Sample taken predose, 1, 3, 5, 7, 9, 13, 18, 24, 36, 48, 72, 96, 144, 216 hours postdose
Description of the pharmacokinetic(PK) profile for in terms of the regression coefficient for calculation of the terminal rate constant (Rsq), and the percentage of area under the curve to infinity obtained by extrapolation (%AUCex). | Sample taken predose, 1, 3, 5, 7, 9, 13, 18, 24, 36, 48, 72, 96, 144, 216 hours postdose
Description of the pharmacokinetic(PK) profile for in terms of the metabolic ratios (ratio of metabolite to parent) for AUC and Cmax (MRAUC and MRCmax) | Sample taken predose, 1, 3, 5, 7, 9, 13, 18, 24, 36, 48, 72, 96, 144, 216 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: James Ritter, MD, Principal Investigator — Quintiles London UK; Bengt Larsson, MD, Study Director — Astrazeneca Molndal, Sweden; Stuart Oliver, MD, Study Chair — Astrazeneca UK
Locations (1):
- Research Site, London, United Kingdom

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1848&filename=D5200C00001_Study_Synopsis.pdf